CLINICAL TRIAL: NCT04758845
Title: A Randomized, 5 Arm, Parallel, Placebo Controlled Clinical Study to Evaluate Safety and Efficacy of New Probiotic Strains in Healthy Adults
Brief Title: Clinical Study to Evaluate the Safety and Efficacy of New Probiotic Strains in Health Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deerland Enzymes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pro5Safe
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Gastrointestinal Health; Respiratory Health; Safety
Keywords: Probiotics; Gastrointestinal Health; Respiratory Health; Immunomodulation; Antioxidant; Chelation of heavy metals

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cocktail (Experimental): Subjects will consume 1 capsule containing 2B CFU containing .5B CFU Bacillus subtilis DE111, .5B CFU Bacillus coagulans CGI314, .5B CFU Bacillus megaterium MIT411, and .5B CFU Bacillus clausii CSI08 for 45 days.
  Interventions: Dietary Supplement: Cocktail
- CGI314 (Experimental): Subjects will consume 1 capsule containing 1B CFU of Bacillus coagulans CGI314 for 45 days.
  Interventions: Dietary Supplement: CGI314
- CSI08 (Experimental): Subjects will consume 1 capsule containing 1B CFU of Bacillus clausiiCSI08 for 45 days.
  Interventions: Dietary Supplement: CSI08
- MIT411 (Experimental): Subjects will consume 1 capsule containing 1B CFU of Bacillus megaterium MIT411 for 45 days.
  Interventions: Dietary Supplement: MIT411
- Placebo (No Intervention): Subjects will consume 1 capsule containing maltodextrin for 45 days.

INTERVENTIONS:
Dietary Supplement: Cocktail — Subjects will consume 2B CFU once daily containing .5B CFU DE111, .5B CFU MIT411, .5B CFU CGI314, and .5B CFU CSI08 for 45 days.
  Arms: Cocktail
Dietary Supplement: CGI314 — Subjects will consume 1B CFU of CGI314 once daily for 45 days.
  Arms: CGI314
Dietary Supplement: CSI08 — Subjects will consume 1B CFU of CSI08 once daily for 45 days.
  Arms: CSI08
Dietary Supplement: MIT411 — Subjects will consume 1B CFU of MIT411 once daily for 45 days.
  Arms: MIT411

SUMMARY:
This trial is to determine the safety of 4 new probiotic strains and to assess their efficacy in reducing the incidence and/or duration of gastrointestinal problems and infections as well as respiratory infections in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form. Healthy adults aged 18-65.

Exclusion Criteria:

* Presence of a pre-existing adverse events monitored in the study. Presence of a serious congenital anomaly or chronic medical condition that would contraindicate participation, including history of major GI surgery, chronic GI illness, abnormal intestinal anatomy or significant abdominal disorder. Severe chronic illness. Known immunodeficiency. Use of immunosuppressive agents. Presence of severe immunodeficient family members. Pregnancy, 6 months postpartum period or currently breastfeeding. Women of child bearing age planning pregnancy during the course of the study. Participation in another study. Not able to understand and comply with requirements of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Safety | 45 days
  Participants will be asked to note any adverse events that might occur during 45 days study treatment period in the participant diary 1 and 14 days follow-up period in the participant diary 2 and to call the investigator if any clinically significant events occur. The investigator will review the returned participant diaries together with the participant. Based on the adverse events marked in the diaries and written in medical records the number of adverse event occurrences, their nature and causality will be evaluated in all study regimes.

SECONDARY OUTCOMES:
Immunomodulation | 45 days
  Evaluate difference in salivary IgA in experimental groups compared to placebo
Regularity | 45 days
  Evaluate difference in stool consistency according to Bristol stool chart, and regularity of defecation from baseline to day 45 in experimental groups compared to control group and from baseline to end of 14 days follow up period (59 days) in the experimental groups compared to control group. Participants will be asked to track the type of their stool using the bristol stool chart, and times of defecation during the 45 day treatment period and 14 days follow up period in their diaries. On visit 2 and during the follow up phone call the investigator will review the participant diary together with the participant.
GI Health | 45 days
  Assess number of days with gastrointestinal problems in experimental groups compared to placebo.
Respiratory Health | 45 days
  Assess number of days with respiratory infections in experimental groups compared to placebo.

OTHER OUTCOMES:
Heart Health | 45 days
  Assess the change in blood lipids from baseline to finish in experimental groups compared to plcaebo
Inflammation | 45 days
  Assess the change in cytokines in experimental groups compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Lilijana K Besednjak, MD PhD, Principal Investigator — Health Center Nova Gorica
Locations (1):
- Health Center Nova Gorica, Šempeter pri Gorici, Slovenia

REFERENCES:
- [Derived] Rea K, Colom J, Simon EA, Khokhlova E, Mazhar S, Barrena M, Enrique M, Martorell P, Perez BA, Tortajada M, Phipps C, Deaton J. Evaluation of Bacillus clausii CSI08, Bacillus megaterium MIT411 and a Bacillus cocktail on gastrointestinal health: a randomised, double-blind, placebo-controlled pilot study. Benef Microbes. 2023 Apr 18;14(2):165-182. doi: 10.3920/BM2022.0117. Epub 2023 Apr 7. PMID 37026366